CLINICAL TRIAL: NCT02225119
Title: The Focal Electro-Oculogram in Macular Disease
Status: Completed | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 140171; 14-EI-0171
Record Dates: First submitted 2014-08-23; First posted 2014-08-26 (Estimated); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Macular Degeneration; Age-Related Macular Degeneration
Keywords: Retinal Images; Retinal Pigment Epithelium; Natural History
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Affected: Participants with macular disease
- Unaffected: Healthy volunteers

SUMMARY:
Background:

- Maculopathies are eye conditions that affect the center of the retina. Retina health depends on the retinal pigment epithelium (RPE), a layer behind the retina. A new test may measure the health of the central retina and RPE.

Objective:

- To use the focal electro-oculogram (EOG) test to understand how the central retina and RPE are affected in maculopathies.

Eligibility:

* People at least 10 years old with a maculopathy.
* Healthy volunteers with visual acuity of 20/20 or better in at least one eye.

Design:

* Participants will be screened with medical and eye history and an eye exam. Pictures will be taken of the eyes.
* Their eyes may be dilated.
* They may have a field test. They will look into a lens and press a button when they see a light. First, they may sit in the dark for 40 minutes.
* Participants will have 1-7 visits over 18 months.
* Their vision will be tested and eye pressure measured.
* Their pupils will be dilated with eye drops and researchers may take pictures of the retina and the inside of the eye, and measure the thickness of the retina.
* Participants will have an electro-oculogram. They will look at a 2 LED lights and follow them back and forth for 10 seconds once per minute. Participants will be in darkness for 15 minutes and in light for 20 minutes. One skin electrode will be placed on the nose and one next to the eye.
* Participants with maculopathy will also have:
* Field test.
* Electroretinogram. Participants will get numbing eye drops and special contact lenses. A small metal electrode will be taped to the forehead. Participants will watch flashing lights and try not to blink. First, they may sit in the dark for 40 minutes.

DETAILED DESCRIPTION:
OBJECTIVE:

The objective of this protocol is to investigate the local response of the retinal pigment epithelium (RPE) across the posterior pole of the eye by recording the focal electrooculogram (EOG) in participants with macular disease.

STUDY POPULATION:

Up to 50 healthy volunteers and 80 participants, age 10 or older, with macular disorders affecting the retina/retinal pigment epithelium complex. Examples of such macular disorders include Stargardt s disease and age-related macular degeneration (AMD).

DESIGN:

This single-center, observational, case-control study will be comprised of three related aims. The first aim is focused on developing the focal EOG method which will require parameter optimization. The second aim is focused on establishing the normal range and variability of the focal EOG in normal volunteers. The third aim is to examine the focal EOG in participants with macular disease.

OUTCOME MEASURES:

The primary outcome for this study is to develop a method for recording the focal EOG. The secondary outcome will be to establish the normal range for the focal EOG and determine the inter-session and intra-session variabilities of this test. Exploratory outcomes include: 1) to examine the focal EOG in participants with macular diseases and 2) determine the inter-session and intra-session variabilities of this test in participants with macular diseases.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Participant must be 10 years of age or older.
  2. Participant (or legal guardian) must understand and sign the protocol s informed consent document.
  3. Participant must be able to cooperate with the testing required for this study.
  4. For Participants with macular disease only:

     1. Participant must have macular disease, defined as evidence of loss of centrally mediated retinal dysfunction and/or degeneration as established by standard clinical methods including perimetry, ERG and imaging.
     2. Participant must have a measurable visual acuity.
  5. For Healthy Volunteers only:

     1. Participant must have visual acuity of 20/20 or better in at least one eye.

EXCLUSION CRITERIA:

1) Participant with pre-retinal media opacities that would prevent focal light presentation.

Ages: 10 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Up to 50 healthy volunteers and 80 participants, age 10 or older, with macular disease; examples of such disorders include Stargardt s disease and age-related macular degeneration (AMD). NIH employees meeting the eligibility criteria may participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2015-02-06 (Actual); Primary Completion 2019-05-07 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
develop method for recording focal EOG | up to 6 months
  to develop a method for recording the focal EOG in response to a central light stimulus

SECONDARY OUTCOMES:
establish the normal range for the focal EOG and determine the inter-session and intra-session variabilities of this test | up to 18 months
  establish the normal range for the focal EOG and determine the inter-session and intra-session variabilities of this test

CONTACTS AND LOCATIONS:
Overall Officials: Brett G Jeffrey, Ph.D., Principal Investigator — National Eye Institute (NEI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2014-EI-0171.html